CLINICAL TRIAL: NCT07232953
Title: Prospective Phase II Study on Safety and Efficacy of Fludarabine Plus Treosulfan (14g) (FT14) Conditioning Regimen for Allogeneic Stem Cell Transplantation (Allo-SCT) in Acute Myeloid Leukemia (AML) Patients (≥40 <65years) (FT14-Trial)
Brief Title: Safety and Efficacy of FT14 Conditioning for Allogeneic HSCT in Acute Myeloid Leukemia
Acronym: FT14
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Prof Domenico Russo, Principal Investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT14-Trial
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukaemia (AML); Hematopoietic Stem Cell Transplant (HSCT)
Keywords: AML; Fludarabine; Treosulfan; Allo-HSCT
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; treosulfan

STUDY DESIGN:
Intervention Model Description: This is a multicenter, non-randomized, open-label, single-arm phase II study in which all enrolled patients receive the same conditioning regimen with Fludarabine plus Treosulfan (FT14) before allogeneic stem cell transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fludarabine + Treosulfan conditioning regimen in AML patients (Experimental): Fludarabine (30 mg/m²/d × 5 days) IV infusion days -6 to -2 and Treosulfan (14 g/m²/d × 3 days) IV infusion days -4 to -2.
  Interventions: Drug: Fludarabine + Treosulfan

INTERVENTIONS:
Drug: Fludarabine + Treosulfan — Fludarabine (30 mg/m²/d × 5 days) IV infusion days -6 to -2 and Treosulfan (14 g/m²/d × 3 days) IV infusion days -4 to -2
  Other Names: Treosulfan; Fludarabine

SUMMARY:
This is a prospective, multicenter, phase II, open-label, non-randomized clinical trial designed to evaluate the safety and efficacy of the Fludarabine plus Treosulfan 14 g/m² (FT14) conditioning regimen for allogeneic stem cell transplantation (allo-SCT) in patients with Acute Myeloid Leukemia (AML) aged 40-65 years who are in complete remission.

DETAILED DESCRIPTION:
This is a prospective, multicenter, phase II, open-label, non-randomized clinical trial designed to evaluate the safety, tolerability, and antileukemic activity of the FT14 conditioning regimen (Fludarabine plus Treosulfan 14 g/m²/day for three consecutive days) in adult patients with Acute Myeloid Leukemia (AML) undergoing allogeneic hematopoietic stem cell transplantation (allo-HSCT). Eligible patients are 40 to 65 years old, in complete remission (CR), and candidates for allogeneic transplantation according to institutional criteria.

Treosulfan-based conditioning represents an effective alternative to conventional myeloablative regimens, with reduced organ toxicity and favorable immunosuppressive properties. Increasing the treosulfan dose to 14 g/m²/day aims to enhance antileukemic potency while maintaining an acceptable safety profile. Fludarabine provides additional immunosuppression and cytotoxic synergism, facilitating engraftment and disease control.

Enrolled patients will receive the FT14 conditioning regimen followed by allo-HSCT from either a matched related donor (MRD) or a matched unrelated donor (MUD). Haploidentical donors are not included in this study. Graft-versus-host disease (GVHD) prophylaxis, antimicrobial prophylaxis, and supportive care will follow each center's standard procedures.

The primary endpoint is the 1-year leukemia-free survival (LFS). Secondary endpoints include time to engraftment, cumulative incidence of graft failure, transplant-related mortality (TRM) and non-relapse mortality (NRM), relapse incidence, acute and chronic GVHD incidence and severity, overall survival (OS), and graft-versus-host disease-free, relapse-free survival (GRFS). Safety will be assessed through regimen-related toxicities, early and late post-transplant complications, and hematologic recovery kinetics.

The study is designed to provide prospective clinical evidence on the performance, tolerability, and efficacy of the FT14 regimen in adults with AML undergoing allo-HSCT, with the aim of defining its potential role as a conditioning option for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients >40 <65 years of age
* Diagnosis of AML in first complete remission (CR)/complete remission with incomplete recovery (CRi)/multiflow leukemia free state (MLFS)
* Eligible for allo-SCT from HLA-identical matched related or unrelated donor as defined by molecular high-resolution typing (4 digits) at the following four HLA gene loci (HLA-A, B, C, and DRB1)
* Adequate hepatic function (bilirubin ≤2 UNL; ALT/AST ≤2,5 UNL)
* Adequate renal function (creatinine clearance ≥50 mL/min)
* ECOG Performance Status < 2
* Willing and able to comply with all of the requirements and visits in the protocol.
* Written and signed informed consent

Exclusion Criteria:

* AML patients with t(15;17); t(8;21); inv(16)
* Subject has known active CNS involvement with AML.
* Grade >2 NCI-CTCAE (v. 5) adverse events at the time of enrollment
* Serious organ dysfunction: left ventricular ejection fraction < 40%, FEV1, FVC, DLCO (diffusion capacity) <40% of predicted, LFT > 5 times the upper limit of normal, or creatinine clearance < 40 ml/min.
* The evidence of HBV or HCV active infection (HBV DNA, HCV RNA positive test).
* Patients with HIV infection
* Current uncontrolled infections
* Patients with other life-threatening concurrent diseases
* Subjects with known hypersensitivity to any of the component medications
* Participation in another clinical trial within 1 month before the start of this trial
* Participant, both female and male, in childbearing age who do not agree to maintain an active contraceptive practice
* Pregnant or breastfeeding patients during screening

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The 1-year leukemia -free survival (LFS) after allo-SCT | From allo-HSCT to 1-year post allo-HSCT
  Proportion of patients alive and free from leukemia at 1 year after allogeneic hematopoietic stem cell transplantation (allo-HSCT), estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Cumulative incidence of graft failure at day +30 | From allo-HSCT to day +30
  Cumulative incidence of primary graft failure within 30 days after allo-HSCT, considering death without graft failure as a competing risk.
Cumulative incidence of graft failure at day +100 | From allo-HSCT to day +100
  Cumulative incidence of primary or secondary graft failure within 100 days after allo-HSCT, with competing-risk methodology.
Transplant-related mortality (TRM) at day +100 | From allo-HSCT to day +100
  Proportion of patients who die without evidence of disease relapse within 100 days after allo-HSCT (non-relapse mortality), estimated using cumulative incidence.
TRM at 1 year | From allo-HSCT to 1 year
  Cumulative incidence of TRM within 1 years after allo-HSCT.
TRM at 2 years | From allo-HSCT to 2 years
  Cumulative incidence of TRM within 2 years after allo-HSCT.
Cumulative incidence of acute GVHD at day +100 | From allo-HSCT to day +100
  Proportion of patients developing grade II-IV acute GVHD by day +100, estimated using cumulative incidence with relapse and death as competing events.
Cumulative incidence of chronic GVHD at 1 year | From allo-HSCT to 1 year
  Cumulative incidence of chronic GVHD diagnosed within 1 year after allo-HSCT, based on NIH criteria, using competing-risk methodology.
Cumulative incidence of chronic GVHD at 2 years | From allo-HSCT to 2 years
  Cumulative incidence of chronic GVHD diagnosed within 2 years after allo-HSCT, based on NIH criteria.
Relapse incidence at 1 year | From allo-HSCT to 1 year
  Cumulative incidence of leukemia relapse within 1 year after allo-HSCT, analyzed using competing-risk models.
Relapse incidence at 2 year | From allo-HSCT to 2 year
  Cumulative incidence of leukemia relapse within 2 year after allo-HSCT, analyzed using competing-risk models.
Overall survival at 1 year | From allo-HSCT to 1 year
  Proportion of patients alive at 1 year after allo-HSCT, estimated by Kaplan-Meier analysis.
Overall survival at 2 years | From allo-HSCT to 2 years
  Proportion of patients alive at 2 years after allo-HSCT, estimated by Kaplan-Meier method.
Graft-versus-Host Disease-Free, Relapse-Free Survival (GRFS) at 1 year | From allo-HSCT to 1 year
  Proportion of patients alive without grade III-IV acute GVHD, chronic GVHD requiring systemic therapy, relapse, or death at 1 year after allo-HSCT.
GRFS at 2 years | From allo-HSCT to 2 years
  Proportion of patients alive without severe acute GVHD, chronic GVHD requiring systemic therapy, relapse, or death within 2 years after allo-HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Russo, MD, Principal Investigator — ASST Spedali Civili di Brescia
Locations (13):
- Italy (13):
  - Grande Ospedale Metropolitano "Bianco Melacrino Morelli", Reggio Calabria, Calabria
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli, Napoli, Campania
  - Azienda Ospedaliera Universitaria di Modena, Modena, Emilia-Romagna
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine, Friuli Venezia Giulia
  - ASST degli Spedali Civili di Brescia, Brescia, Lombardy
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico,, Milan, Lombardy
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Azienda Ospedaliera S. Croce e Carle, Cuneo, Piedmont
  - Ospedali Riuniti di Ancona, Ancona, The Marches
  - Ospedale C e G Mazzoni, Ascoli Piceno, The Marches
  - Azienda Ospedaliero Universitaria Careggi, Florence, Tuscany
  - Ospedale dell'Angelo, Mestre, Veneto
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona, Veneto

IPD SHARING:
Plan to Share IPD: No
At this time, individual participant data will not be shared outside the study team.

REFERENCES:
- [Result] Shimoni A, Labopin M, Savani B, Hamladji RM, Beelen D, Mufti G, Socie G, Delage J, Blaise D, Chevallier P, Forcade E, Deconinck E, Mohty M, Nagler A. Intravenous Busulfan Compared with Treosulfan-Based Conditioning for Allogeneic Stem Cell Transplantation in Acute Myeloid Leukemia: A Study on Behalf of the Acute Leukemia Working Party of European Society for Blood and Marrow Transplantation. Biol Blood Marrow Transplant. 2018 Apr;24(4):751-757. doi: 10.1016/j.bbmt.2017.12.776. Epub 2017 Dec 13. PMID 29247780
- [Result] Ruutu T, Volin L, Beelen DW, Trenschel R, Finke J, Schnitzler M, Holowiecki J, Giebel S, Markiewicz M, Uharek L, Blau IW, Kienast J, Stelljes M, Larsson K, Zander AR, Gramatzki M, Repp R, Einsele H, Stuhler G, Baumgart J, Mylius HA, Pichlmeier U, Freund M, Casper J. Reduced-toxicity conditioning with treosulfan and fludarabine in allogeneic hematopoietic stem cell transplantation for myelodysplastic syndromes: final results of an international prospective phase II trial. Haematologica. 2011 Sep;96(9):1344-50. doi: 10.3324/haematol.2011.043810. Epub 2011 Jun 9. PMID 21659356
- [Result] Casper J, Holowiecki J, Trenschel R, Wandt H, Schaefer-Eckart K, Ruutu T, Volin L, Einsele H, Stuhler G, Uharek L, Blau I, Bornhaeuser M, Zander AR, Larsson K, Markiewicz M, Giebel S, Kruzel T, Mylius HA, Baumgart J, Pichlmeier U, Freund M, Beelen DW. Allogeneic hematopoietic SCT in patients with AML following treosulfan/fludarabine conditioning. Bone Marrow Transplant. 2012 Sep;47(9):1171-7. doi: 10.1038/bmt.2011.242. Epub 2011 Dec 12. PMID 22158386
- [Result] Westerhof GR, Ploemacher RE, Boudewijn A, Blokland I, Dillingh JH, McGown AT, Hadfield JA, Dawson MJ, Down JD. Comparison of different busulfan analogues for depletion of hematopoietic stem cells and promotion of donor-type chimerism in murine bone marrow transplant recipients. Cancer Res. 2000 Oct 1;60(19):5470-8. PMID 11034090
- [Result] Fichtner I, Becker M, Baumgart J. Antileukaemic activity of treosulfan in xenografted human acute lymphoblastic leukaemias (ALL). Eur J Cancer. 2003 Apr;39(6):801-7. doi: 10.1016/s0959-8049(02)00767-0. PMID 12651206
- [Result] Munkelt D, Koehl U, Kloess S, Zimmermann SY, Kalaaoui RE, Wehner S, Schwabe D, Lehrnbecher T, Schubert R, Kreuter J, Klingebiel T, Esser R. Cytotoxic effects of treosulfan and busulfan against leukemic cells of pediatric patients. Cancer Chemother Pharmacol. 2008 Oct;62(5):821-30. doi: 10.1007/s00280-007-0669-3. Epub 2008 Feb 2. PMID 18246351
- [Result] Beelen DW, Trenschel R, Stelljes M, Groth C, Masszi T, Remenyi P, Wagner-Drouet EM, Hauptrock B, Dreger P, Luft T, Bethge W, Vogel W, Ciceri F, Peccatori J, Stolzel F, Schetelig J, Junghanss C, Grosse-Thie C, Michallet M, Labussiere-Wallet H, Schaefer-Eckart K, Dressler S, Grigoleit GU, Mielke S, Scheid C, Holtick U, Patriarca F, Medeot M, Rambaldi A, Mico MC, Niederwieser D, Franke GN, Hilgendorf I, Winkelmann NR, Russo D, Socie G, Peffault de Latour R, Holler E, Wolff D, Glass B, Casper J, Wulf G, Menzel H, Basara N, Bieniaszewska M, Stuhler G, Verbeek M, Grass S, Iori AP, Finke J, Benedetti F, Pichlmeier U, Hemmelmann C, Tribanek M, Klein A, Mylius HA, Baumgart J, Dzierzak-Mietla M, Markiewicz M. Treosulfan or busulfan plus fludarabine as conditioning treatment before allogeneic haemopoietic stem cell transplantation for older patients with acute myeloid leukaemia or myelodysplastic syndrome (MC-FludT.14/L): a randomised, non-inferiority, phase 3 trial. Lancet Haematol. 2020 Jan;7(1):e28-e39. doi: 10.1016/S2352-3026(19)30157-7. Epub 2019 Oct 9. PMID 31606445
- [Result] Romanski M, Wachowiak J, Glowka FK. Treosulfan Pharmacokinetics and its Variability in Pediatric and Adult Patients Undergoing Conditioning Prior to Hematopoietic Stem Cell Transplantation: Current State of the Art, In-Depth Analysis, and Perspectives. Clin Pharmacokinet. 2018 Oct;57(10):1255-1265. doi: 10.1007/s40262-018-0647-4. PMID 29557088
- [Result] Danylesko I, Shimoni A, Nagler A. Treosulfan-based conditioning before hematopoietic SCT: more than a BU look-alike. Bone Marrow Transplant. 2012 Jan;47(1):5-14. doi: 10.1038/bmt.2011.88. Epub 2011 Apr 11. PMID 21478921
- [Result] Rambaldi A, Grassi A, Masciulli A, Boschini C, Mico MC, Busca A, Bruno B, Cavattoni I, Santarone S, Raimondi R, Montanari M, Milone G, Chiusolo P, Pastore D, Guidi S, Patriarca F, Risitano AM, Saporiti G, Pini M, Terruzzi E, Arcese W, Marotta G, Carella AM, Nagler A, Russo D, Corradini P, Alessandrino EP, Torelli GF, Scime R, Mordini N, Oldani E, Marfisi RM, Bacigalupo A, Bosi A. Busulfan plus cyclophosphamide versus busulfan plus fludarabine as a preparative regimen for allogeneic haemopoietic stem-cell transplantation in patients with acute myeloid leukaemia: an open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2015 Nov;16(15):1525-1536. doi: 10.1016/S1470-2045(15)00200-4. Epub 2015 Sep 28. PMID 26429297
- [Result] Rashidi A, Weisdorf DJ, Bejanyan N. Treatment of relapsed/refractory acute myeloid leukaemia in adults. Br J Haematol. 2018 Apr;181(1):27-37. doi: 10.1111/bjh.15077. Epub 2018 Jan 9. PMID 29318584